CLINICAL TRIAL: NCT00823043
Title: A Comfort Survey of Open-angle Glaucoma or Ocular Hypertension Patients Treated With Timolol Hemihydrate 0.5% Solution Once or Twice Daily Versus Timolol Maleate in Sorbate
Brief Title: A Comfort Survey of Open-angle Glaucoma or Ocular Hypertension Patients Treated With 2 Drugs
Status: Completed | Type: Observational
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VPH0110
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Timolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Timolol hemihydrate: Subjects currently prescribed timolol hemihydrate 0.5% solution.
  Interventions: Drug: timolol hemihydrate
- Timolol maleate: Subjects currently prescribed timolol maleate in sorbate.
  Interventions: Drug: timolol maleate

INTERVENTIONS:
Drug: timolol hemihydrate — timolol hemihydrate 0.5% solution
  Groups: Timolol hemihydrate
Drug: timolol maleate — timolol maleate in sorbate
  Groups: Timolol maleate

SUMMARY:
The objective of the study was to evaluate whether timolol hemihydrate is more comfortable upon instillation than timolol maleate in sorbate. This was an observational study. Subjects with open-angle glaucoma or ocular hypertension were asked to complete a survey regarding their normal treatment. No treatment was prescribed.

ELIGIBILITY:
Inclusion Criteria:

* willing to comply with investigator's and protocol's instructions
* patients signature on the informed consent document
* open-angle glaucoma or ocular hypertension
* currently prescribed timolol hemihydrate (once a day (QD) or twice a day (BID))or timolol maleate in sorbate QD as monotherapy or as a part of 2-drug therapy in at least one eye

Exclusion Criteria:

* inability to understand the trial procedures
* inability to give informed consent
* inability to understand, read, or write English
* best corrected visual acuity of 20/200 or worse in each eye
* current moderate to severe infectious or inflammatory condition of the eye or eyelids including
* current moderate to severe dry eye syndrome
* current chronic use of ocular corticosteroids, ocular surgery or intraocular laser surgery to either eye in the prior 3 months
* treated with 3 or more glaucoma medicines in both eye

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in centers in the United States with substantial populations of patients prescribed timolol hemihydrate and timilol maleate in sorbate.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — PRN Pharmacuetical Research Network, LLC
Locations (1):
- Eye Care of San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Timolol Hemihydrate: Timolol hemihydrate 0.5% ophthalmic solution.
- Timolol Maleate in Sorbate: Timolol maleate in sorbate 0.5% ophthalmic solution
Period: Overall Study
Arm/Group | Timolol Hemihydrate | Timolol Maleate in Sorbate
Started | 64 | 39
Completed | 64 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Subject Population: All subjects responding to survey
Arm/Group | Total Subject Population
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Burning/Stinging
Description: Subjects reported burning/stinging after they put the drops in their eyes using the following scale: 0=never, 1=rarely, 2=sometimes, 3=frequently, 4=always.
Time Frame: Upon instillation
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Timolol Hemihydrate | Timolol Maleate in Sorbate
Number analyzed (Participants) | 64 | 39
Units on a Scale | 1.1 (1.1) | 2.4 (1.4)
Statistical Analysis 1: Comparison: Timolol Hemihydrate vs Timolol Maleate in Sorbate; Test type: Superiority or Other; p < .001, t-test, 2 sided

2. Primary Outcome: Subject Reported Tearing
Description: Subjects reported tearing after they put the drops in their eyes using the following scale:0=never, 1=rarely, 2=sometimes, 3=frequently, 4=always.
Time Frame: Upon instillation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Timolol Hemihydrate | Timolol Maleate in Sorbate
Number analyzed (Participants) | 64 | 39
Units on a Scale | 0.9 (1.0) | 1.6 (1.6)
Statistical Analysis 1: Comparison: Timolol Hemihydrate vs Timolol Maleate in Sorbate; Test type: Superiority or Other; p = 0.024, t-test, 2 sided

3. Primary Outcome: Subject Reported Light Sensitivity
Description: Subjects reported light hurt their eyes after they put the drops in their eyes using the following scale: 0=never, 1=rarely, 2=sometimes, 3=frequently, 4=always.
Time Frame: Upon instillation
Population: Analysis includes all subjects that answered this question. One subject from each arm did not answer this question.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Timolol Hemihydrate | Timolol Maleate in Sorbate
Number analyzed (Participants) | 63 | 38
Units on a Scale | 0.5 (0.7) | 0.4 (0.9)
Statistical Analysis 1: Comparison: Timolol Hemihydrate vs Timolol Maleate in Sorbate; Test type: Superiority or Other; p = 0.75, t-test, 2 sided

4. Primary Outcome: Subject Reported Blurred Vision
Description: Subjects reported their vision was blurred after they put the drops in their eyes using the following scale: 0=never, 1=rarely, 2=sometimes, 3=frequently, 4=always.
Time Frame: Upon instillation
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Timolol Hemihydrate | Timolol Maleate in Sorbate
Number analyzed (Participants) | 64 | 39
Units on a Scale | 0.7 (1.0) | 0.6 (1.0)
Statistical Analysis 1: Comparison: Timolol Hemihydrate vs Timolol Maleate in Sorbate; Test type: Superiority or Other; p = 0.69, t-test, 2 sided

ADVERSE EVENTS:
Description: This was an observational study. Subjects with open-angle glaucoma or ocular hypertension were asked to complete a survey regarding their normal treatment. No treatment was prescribed and adverse event questions were not included in the survey.
Arm/Group | Total Subjects Surveyed
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the PI will provide the Sponsor with at least 60 days for review of a manuscript. If requested in writing, the PI will withhold publication for up to an additional 60 days.